CLINICAL TRIAL: NCT01852617
Title: A Smoking Cessation Intervention During Pregnancy in Argentina and Uruguay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Tulane University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ezequiel Garcia Elorrio, Chief of Administration, Institute for Clinical Effectiveness and Health Policy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1U48DP001948-01 (NIH)
Record Dates: First submitted 2011-06-22; First posted 2013-05-14 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Smoking Cessation; Pregnancy
Keywords: Smoking Cessation; Pregnancy; Implementation; Knowledge translation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation of intervention (Experimental): Midwife facilitators in the intervention clinics will be identified and trained to deliver the "5 A's" to pregnant women and will then disseminate and implement the program. The "5 A's" (Ask, Advise, Assess, Assist, Arrange) is a strategy consisting of a brief cessation counseling session of 5-15 minutes delivered by a trained provider, which is considered the standard of care worldwide
  Interventions: Behavioral: Training in smoking cessation counseling
- No implementation of the intervention (No Intervention): Standard in-service activities

INTERVENTIONS:
Behavioral: Training in smoking cessation counseling — Midwife facilitators in the intervention clinics will be identified and trained to deliver the "5 A's" to pregnant women and will then disseminate and implement the program. The "5 A's" (Ask, Advise, Assess, Assist, Arrange) is a strategy consisting of a brief cessation counseling session of 5-15 minutes delivered by a trained provider, which is considered the standard of care worldwide
  Arms: Implementation of intervention

SUMMARY:
Argentina and Uruguay are among the countries with the highest proportion of pregnant women who smoke. The implementation of an effective smoking cessation intervention would have a significant impact on the health of mothers and children. The "5 A's" (Ask, Advise, Assess, Assist, Arrange) is a strategy consisting of a brief cessation counseling session of 5-15 minutes delivered by a trained provider, which is considered the standard of care worldwide. However, it is under used in Argentina and Uruguay. We will conduct a two-arm, parallel cluster randomized controlled trial of an implementation intervention in 20 prenatal clinics in Argentina and Uruguay. Our primary hypothesis is that the intervention is feasible in prenatal clinics in Argentina and Uruguay and will increase the frequency of women receiving tobacco use cessation counseling during pregnancy. Our secondary hypothesis is that the intervention will decrease the frequency of women who smoke by the end of their pregnancies. Prenatal clinics will be randomly allocated to either an intervention or a control group after a baseline data collection period. Midwife facilitators in the ten intervention clinics will be identified and trained to deliver the "5 A's" to pregnant women and will then disseminate and implement the program. The ten clinics in the control group will continue with their standard in-service activities. A follow-up data collection will be conducted immediately after delivery. The intervention will be tailored by formative research to be readily applicable to local prenatal care services at busy maternity hospitals, as well as to be acceptable to local pregnant women and health providers. The study will be conducted in 48 months.

ELIGIBILITY:
Inclusion Criteria por prenatal clinics:

* Not having a smoking cessation program based on the "5 A's" for pregnant women in place.
* An estimated frequency of women receiving the "5 A's" intervention below 20%
* Having midwives or nurse-midwives as part of the hospital or primary health center staff.
* Having signed a letter of intention to participate in the project.
* Having at least 400 new pregnant women per year.

Exclusion Criteria for prenatal clinics:

* None

Ages: 12 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6858 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Frequency of women receiving the cessation smoking advice | Interviews during the first 12 hours after delivery
  Frequency of women receiving the "5 A's" (ask smoking status of all women; advise smokers to quit; assess their willingness to make a quit attempt; assist their attempt by providing skills and materials for tobacco cessation; arrange: monitor smoking status at all prenatal visits) in women having prenatal care at the participating prenatal clinics.

SECONDARY OUTCOMES:
Frequency of women who smoke at the end of pregnancy | Interviews and saliva samples during the first 12 hours after delivery
  Frequency of women who smoke at the end of pregnancy: Women will be interviewed during their postpartum hospital stay and saliva samples will be taken for cotinine analysis.
Frequency of providers' positives attitudes and readiness to change | 6 months before and after the implementation of the intervention
  Frequency of positives attitudes and readiness to provide counseling for smoking cessation to women following the "5 A's" model among midwives working at participating prenatal clinics. Assessed through a self-administered questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Althabe, MD, Principal Investigator — Institute for Clinical Effectiveness and Health Policy
Locations (22):
- Argentina (10):
  - Hospital Lucio Meléndez, Adrogué, Buenos Aires
  - Hospital Evita Pueblo, Berazategui, Buenos Aires
  - Hospital M.V de Martínez, General Pacheco, Buenos Aires
  - Hospital Narciso López, Lanús, Buenos Aires
  - Hospital Héroes de Malvinas, Merlo, Buenos Aires
  - Hospital Municipal Ostaciana B. de Lavignolle, Morón, Buenos Aires
  - Hospital Materno Infantil de San Isidro, San Isidro, Buenos Aires
  - Hospital Bocalandro, Tres de Febrero, Buenos Aires
  - Hospital Maternidad Santa Rosa, Vicente López, Buenos Aires
  - Hospital San Roque, Manuel B. Gonnet, La Plata
- Uruguay (12):
  - Centro de Salud Badano Repetto, Montevideo, Montevideo Department
  - Centro de Salud Cerro, Montevideo, Montevideo Department
  - Centro de Salud Misurraco, Montevideo, Montevideo Department
  - Centro de Salud Saint Bois, Montevideo, Montevideo Department
  - Centro Materno Infantil 1, Montevideo, Montevideo Department
  - Centro Materno Infantil 2, Montevideo, Montevideo Department
  - Centro Materno Infantil 3, Montevideo, Montevideo Department
  - Centro Materno Infantil 4, Montevideo, Montevideo Department
  - Centro Materno Infantil 5, Montevideo, Montevideo Department
  - Centro Materno Infantil 6, Montevideo, Montevideo Department
  - Hospital Canzani, Montevideo, Montevideo Department
  - Hospital Pereira Rossell, Montevideo, Montevideo Department

REFERENCES:
- [Derived] Althabe F, Aleman A, Mazzoni A, Berrueta M, Morello P, Colomar M, Ciganda A, Becu A, Gibbons L, Llambi L, Bittar Gonzalez MG, Tong VT, Farr SL, Smith RA, Dietz PM, Johnson C, Buekens P, Belizan JM. Tobacco cessation intervention for pregnant women in Argentina and Uruguay: study protocol. Reprod Health. 2013 Aug 26;10(1):44. doi: 10.1186/1742-4755-10-44. PMID 23971512